CLINICAL TRIAL: NCT00861549
Title: Bioavailability, Pharmacokinetics and Safety Evaluation of Phencynonate Hydrochloride in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PH-CP005; NCT00766428 (obsolete NCT alias); NCT00926679 (obsolete NCT alias)
Record Dates: First submitted 2009-03-10; First posted 2009-03-13 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Bioavailability; Pharmacokinetics; Safety Evaluation
MeSH Terms: interventions — 3-methyl-3-azabicyclo(3,3,1)nonanyl-9-alpha-yl-alpha-cyclopentyl-alpha-phenyl-alpha-glycolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cohort 1 (Experimental): 1mg / 0.5 tablet
  Interventions: Drug: Phencynonate hydrochloride
- cohort 2 (Experimental): 2mg / 1 tablet; crossover with Phencynonate hydrochloride (2mg/1 tablet) made in China
  Interventions: Drug: Phencynonate hydrochloride
- cohort 3 (Experimental): 4mg / 2 tablets
  Interventions: Drug: Phencynonate hydrochloride

INTERVENTIONS:
Drug: Phencynonate hydrochloride — 2mg/tablet

SUMMARY:
The purpose of this study is to evaluate the bioavailability of two formulations (Taiwan and China mainland) of phencynonate hydrochloride tablets and to generate pharmacokinetic and safety profiles of phencynonate hydrochloride in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated informed consent form.
2. Subjects must be ≧ 18 and ≦ 40 years old, healthy, non-smoking male.
3. Subjects with body weight within ± 20% ideal body weight
4. Subjects with urinalysis data within acceptable range, including pH, blood, glucose and protein
5. Subjects with laboratory evaluations data within acceptable range, including serum chemistry examinations (glucose, total cholesterol, TG, SGOT, SGPT, GSP, alkaline phosphatase, total bilirubin, total protein, albumin, r-GT, BUN, creatinine, uric acid) and hematology (complete blood count and platelets)
6. Subjects with acceptable ECG and chest x-ray

Exclusion Criteria:

1. Subjects had taken any drugs within 14 days prior to screening.
2. Subjects with history of glaucoma
3. Subjects with history of ileus
4. Subjects with history of benign prostate hypertrophy with urine retention
5. Subjects with history of myasthenia gravis
6. Subjects with history of asthma
7. Subject with history of any other medical conditions that, in the opinion of the investigator, compromised subject safety or ability to comply with study procedures
8. Subjects with history of drug or alcohol addiction or abuse within 1 year prior to screening
9. Subjects with hypersensitivity to phencynonate hydrochloride or other drugs with similar chemical structure
10. Subjects had donated blood more than 250 mL within the pervious 3 months prior to study
11. Subjects had received any investigational drugs within 1 month prior to screening

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
PK parameters(1)Cmax,Tmax,Elimination half-life,AUC,Vd/F,Clt/F,MRT,relative BA and percentage of protein binding of plasma PCNH and its metabolite (2) D∞(u)and Clr of urine PCNH and its metabolite | 5 or 10 days
Safety Variables:AE/lab. exam./PE/Vital signs/ECG | 5 to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaoh S Lin, M.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- General Clinical Research Center for New Drug Trial, Tri-Service General Hospital, Taipei, Taiwan